CLINICAL TRIAL: NCT03795311
Title: Phase I / II Study Evaluating the Efficacy and Safety of FOLFIRINOX3 Bevacizumab Treatment in Patients With Colorectal Cancer Who Have Failed With Standard Chemotherapy Protocols (FOLFIRINOX 3)
Brief Title: Evaluation of the Efficacy and the Safety of FOLFIRINOX3 Bevacizumab Treatment in Patients With Colorectal Cancer (FOLFIRINOX 3)
Acronym: FOLFIRINOX3
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLFIRINOX3
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer
Keywords: FOLFIRINOX3 Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of chemotherapy molecules (Experimental): The treatment period is divided into 15-day periods.
  Schema of the administration to the treatments which will proceed in the same way with each cycle:
  Bevacizumab (5 mg/kg; during 30 min) + Oxaliplatine (85 mg/m2, during 2 hours) + Acide folinique (400 mg/m2) or Levofolinate de calcium (200 mg/m2) AND Irinotecan (during 2 hours) + 5-fluorouracile (2400 mg/m2 ; 46 hours) + Irinotecan (1 hour)
  Interventions: Drug: FOLFIRINOX Bevacizumab

INTERVENTIONS:
Drug: FOLFIRINOX Bevacizumab — In phase 1, the goal is to define the DLT (maximum tolerated dose). 3 levels of doses will be evaluated with a different dose of irinotecan in each level.
  * Level -1: Bevacizumab + Oxaliplatine + Acide folinique + Irinotecan: 60mg / m2
  * Level 0: Bevacizumab + Oxaliplatine + Acide folinique +Irinotecan: 70mg / m2
  * Level 1: Bevacizumab + Oxaliplatine + Acide folinique +Irinotecan: 90mg / m2
  The inclusion of patients will start at level 0. Dose-limiting toxicities will be identified during the first 2 cycles.

SUMMARY:
In patients in progression after oxaliplatin and irinotecan, the study FOLFIRINOX 3 proposes to evaluate the interest of modifying the standard pattern of administration of the molecule of irinotecan in order to make it more efficient. In combination with other chemotherapy drugs (5-fluorouracil, oxaliplatin, folinic acid and bevacizumab), irinotecan will be administered at the beginning and end of each cycle of chemotherapy, whereas it is normally administered at one time in the regimen. standard of treatment.

The hypothesis of this study is an increase in the objective response rate at 2 months of 10 to 30% with a scheme by FOLFIRINOX3 - bevacizumab compared to an optimal treatment to date by FOLFIRINOX-bevacizumab.

DETAILED DESCRIPTION:
Primary objective

* Main objective of phase I: To evaluate the acute toxicity of treatment with FOLFIRINOX 3 - bevacizumab
* Main objective of phase II: To evaluate the efficacy of treatment with FOLFIRINOX 3 - bevacizumab in terms of objective response according to the RECIST criteria.

Secondary objectives

* To evaluate the efficacy of treatment with FOLFIRINOX 3 - bevacizumab in terms of objective response according to the criteria of CHOI, progression-free survival (PFS) and overall survival (OS)
* To evaluate the late toxicity of treatment with FOLFIRINOX 3 - bevacizumab
* Evaluate the quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Men or women
2. Age ≥ 18 years
3. Performance status of 0 or 1 (WHO ECOG Index)
4. Patient with metastatic colon cancer
5. History of chemotherapy treatment including oxaliplatin, irinotecan, antiangiogenic (bevacizumab or aflibercept) and anti-EGFR if indicated
6. Patient eligible for treatment with FOLFIRINOX bevacizumab
7. Tumor evaluation (thoraco-abdominopelvic CT scan) performed within 4 weeks before inclusion with at least one measurable lesion according to RECIST criteria 1.1
8. Patient able and able to abide by the protocol throughout the study, including treatment, visits, scheduled examinations and follow-up.
9. Biological values within the following limits:

   * Bilirubinemia ≤ 1.5 times the upper limit of normal (N)
   * ASAT and ALAT ≤ 5 N
   * Creatinine ≤ 1.5 N and creatinine clearance> 60 mlmin
   * Neutrophils ≥ 1.5. 109 / L
   * Platelets ≥ 150. 109 / L
   * Hemoglobin ≥ 9 g / dL (patients can be included even if they have been transfused).
   * Albuminémie≥30g / L
   * Hepatitis B, C and HIV negative serologies
10. Information note given and signed informed consent
11. Patient affiliated to a social security scheme
12. Women must have effective contraception and must have a negative pregnancy test at the time of entry into the study or must no longer be of childbearing age (ie, postmenopausal, after 60 years and no menstruation for ≥1 year without any other medical cause, OR history of hysterectomy, OR history of bilateral oophorectomy),

Exclusion Criteria:

1. Other cancer in the 5 years prior to entry into the trial or concomitant (except in situ cancer of the cervix or basal cell carcinoma of the skin).
2. Presence of cerebral metastasis (s)
3. Prognosis estimated <3 months
4. Presence of a contraindication to bevacizumab (major surgery in the previous 28 days, risk of arterial thrombosis, risk of haemorrhage, deep vein thrombosis without effective anticoagulant therapy or unbalanced anticoagulant therapy)
5. History of grade 4 toxicity to oxaliplatin, irinotecan, 5FU or bevacizumab
6. Persistence of neuropathy greater than a grade 1
7. Hypersensitivity to one of the compounds of the treatments
8. Participation in course or within 30 days prior to entry into the study to another therapeutic trial with an experimental molecule.
9. Demonstration of a DPYD and / or UGT1A1 mutation
10. Unbalanced serious illness, underlying infection that may prevent the patient from receiving treatment
11. Pregnancy (compulsory pregnancy test at baseline), breastfeeding or lack of effective contraception for men and women of childbearing age
12. Psychiatric illness compromising understanding of information or completion of study
13. Patient under tutorship, curatorship or court of justice
14. Inability to sign informed consent or to undergo medical follow-up of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2025-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Acute toxicities as a Measure of treatment specific Safety and Tolerability | each chemotherapy cycle (15 days) up to progression (6 months on average)
  Acute toxicities will be assessed according to the NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Georges François Leclerc, Dijon, France

REFERENCES:
- [Derived] Bellio H, Roussot N, Bertaut A, Hervieu A, Zanetta S, Tharin Z, Vincent J, Bengrine L, Hennequin A, Guion JF, Boudrant A, Collot T, Ghiringhelli F, Fumet JD. FOLFIRINOX-3 plus bevacizumab (bFOLFIRINOX3) in chemo-refractory metastatic colorectal cancer: a multicenter phase II trial. Future Oncol. 2025 Mar;21(6):699-706. doi: 10.1080/14796694.2025.2461446. Epub 2025 Feb 6. PMID 39913183